CLINICAL TRIAL: NCT06810271
Title: Walk It Off! the Influence of Physical Activity Level on the Recovery from Damaging Resistance Exercise
Acronym: WIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: WIO; 00045256 (Other: University of Toronto Health Sciences Research Ethics Board)
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Exercise Induced Muscle Damage; Physical Activity; Inflammation; Exercise Recovery; Skeletal Muscle Damage; Young Adults; Delayed Onset Muscle Soreness (DOMS)
Keywords: Resistance exercise; Exercise induced muscle damage; Ultrasound; Subjective pain; Physical activity
MeSH Terms: conditions — Motor Activity; Inflammation

STUDY DESIGN:
Intervention Model Description: Study includes a behavioural intervention of high and moderate physical activity, modelled by step counts, as a "treatment", or method to improve recovery from the exercise-induced muscle damage intervention occurring in both high and moderate activity phases.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Activity (Experimental): Requires completion of greater than 10,000 steps per day
  Interventions: Behavioral: Eccentric resistance exercise
- Moderate Activity (Experimental): Requires completion of less than 5,000 steps per day
  Interventions: Behavioral: Eccentric resistance exercise

INTERVENTIONS:
Behavioral: Eccentric resistance exercise — 150 maximal, unilateral eccentric contractions of the quadriceps muscles on a computerized dynamometer.

SUMMARY:
After completing novel activity or exercise we may experience exercise-induced muscle damage (EIMD), resulting in a period of reduced muscle function and delayed onset muscle soreness (DOMS). DOMS is characterized by muscle pain and tenderness that typically resolves within a week. While the precise cause of DOMS is unknown, there is growing evidence implicating damage to the connective tissue that surrounds our muscle fibers and is related to a small amount of inflammation. This inflammation is a normal part of our body's ability to recovery from injuries and may be visualized through the use of ultrasound technology. A variety of recovery techniques have been proposed that may help with the recovery of DOMS such as massage and electrical muscle stimulation, but these are not always accessible. Therefore, we are interested in investigating whether the number of daily steps can affect how you experience DOMS.

DETAILED DESCRIPTION:
Skeletal muscle pain and tenderness typically follow an unaccustomed bout of physical activity involving eccentric or lengthening contractions. The intensity of pain peaks between 24 and 72 h following the cessation of activity and subsides completely between 5 and 7 days after exercise. Delayed-onset muscle soreness (DOMS) refers to physical discomfort, while associated impairments to muscle strength and function reflect the occurrence of exercise-induced muscle damage (EIMD). The result is reduced performance and increased likelihood of further injury during the affected period. In beginners, DOMS may also reduce the likelihood of continuing exercise.

Despite its ubiquity in sport and exercise, the precise mechanism of DOMS remains uncertain. Potential mechanisms include EIMD, inflammation, and immune cell infiltration among others. More recently, evidence has emerged suggesting a greater role of intramuscular connective tissue damage in causing DOMS. Following an acute bout of eccentric exercise, the fascial connective tissue exhibits greater swelling than after a concentric exercise. Furthermore, this swelling was correlated with the severity of DOMS. This novel evidence may aid in directing strategies to mitigate the duration and severity of DOMS.

A variety of treatments for DOMS have been explored with varying degrees of efficacy. Massage has been shown to effectively mitigate DOMS following exercise as it passively increases muscle blood flow and reduces muscle oedema. Electrostimulation has also been shown to produce analgesic effects following unaccustomed exercise, although results are inconsistent. Differences in the treatment design may produce discrepant findings with longer duration, lower frequency stimulation alleviating DOMS, in contrast to shorter duration, higher frequency stimulation. Furthermore, lower-intensity longer-duration recovery modalities that promote muscle blood flow may partially ameliorate the ergolytic effects of DOMS. Based on these findings, active recovery consisting of low-intensity exercise following training which facilitates muscle blood flow might be expected to improve recovery from DOMS. However, active recovery strategies such as submaximal cycling or jogging following exercise has little effect on recovery from unaccustomed exercise. While these protocols do promote the muscle blood flow in the days following the bout of exercise, their intensity may be too great to allow for recovery of the muscle while their duration may be too low to produce a sustained effect. It has recently been shown that low daily step counts (<5000/day) can interfere with the normal recovery from aerobic exercise and reduce the normal benefits to metabolism, highlighting that our habitual activity levels might be the most important variable in recovering from and adapting to the stress of exercise. Therefore, the purpose of this study is to investigate the effect of high (>10,000 steps) and moderate (<5,000) daily step counts on recovery from an unaccustomed bout of resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

- Healthy, recreationally active male and female participants (i.e., weekly MET-minutes > 3000 assessed by International Physical Activity Questionnaire).

Not having a health condition that would compromise their ability to safely participate in the strenuous physical activity involved in our study screened for by the get active questionnaire.

Between 18 and 35 years old.

Body mass index (BMI) between 18.5-30

Self-reported not having engaged in resistance exercise and/or lower body plyometrics for at least 3 months prior to the study.

Willing to abide by the compliance rules of this study.

Self-reported regular menstrual cycle (25-35d) within the last 3 months (female participants).

Exclusion Criteria:

Inability to adhere to any of the compliance rules judged by the principal investigator or medical doctor.

Self-reported regular tobacco use.

Regular use of non-steroidal anti-inflammatory drugs (e.g., Advil)

Use of oral contraceptives (female participants).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in maximal muscle strength between physical activity levels | Daily assessment (every 24 hours) across 96 hours post-exercise
  Maximal voluntary isometric and isokinetic contraction assessed by peak torque via computerized dynamometer.

SECONDARY OUTCOMES:
Delayed onset muscle soreness (DOMS) | Daily assessments (every 24 hours) across 96 hours post-exercise
  Assessing DOMS by subjective pain assessments using a 10 centimetre visual analog scale following standardized movements (i.e., descend/ascend stairs, sit-to-stand), where a minimum of "0" reflects no pain, and maximum of "10" reflects the most pain imaginable. Units will be reported to the nearest millimetre.
Change in muscle and fascial connective tissue thickness | Daily assessment (every 24 hours) across 96 hours post-exercise
  Assessing changes in vastus lateralis and rectus femoris muscle and fascial connective tissue thickness via ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Center for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided